

Document Date: 8/22/2022

# Department of Psychiatry and Behavioral Sciences

Box 0984 401 Parnassus Ave. San Francisco, CA 94143

tel: 415.476.7730 fax: 415.476.7320

psychiatry.ucsf.edu

Clinical Trials Official Title: Adapting a Web-Based Professional Development for Mexican School Mental Health Providers Delivering Evidence-Based

Intervention for ADHD and ODD

**Protocol ID: CLSRFUERTE** 

NCT05425966

Principal Investigator: Dr. Lauren M Haack PhD

IRB Study Title: Remote School-Home Program to Improve Youth Attention and

Behavior in Mexican Students

IRB #: 21-34748

**Reference #: 321420** 

Committee of Record: San Francisco General Hospital Panel

**Most Recent Approval Date**: 08/22/2022

Pages 2-35 of the current document: Informed Consent and Assent forms



#### ASSENT TO BE IN A RESEARCH STUDY

# Remote School-Home Program to Improve Youth Attention and Behavior in Mexican Students For children 5 – 12 years old

#### Why are we meeting with you?

We want to tell you about something we are doing called a research study. A research study is when doctors collect a lot of information to learn more about something. Dr. Eva Araujo and some other doctors are doing a study to learn more about how to help children make friends and do better in school. After we tell you about it, we will ask if you'd like to be in this study or not.

#### Why are we doing this study?

We are doing a study that looks at ways to help children. We are hoping to learn more about the kinds of things that might help children do better at school and get along better with other kids and their families. In the whole study, there will be about 88 kids and their families.

### What will happen to you if you are in the study?

If you agree to be in the study, this is what will happen:

We will ask you and your parents and teachers questions about how you are doing at home, at school and with friends.

Then will be in a remote group with other children at your school over videoconferencing. This group will meet 6 times for about one hour each time. You will learn new ways to get along with others, play games, and stay organized. The group is meant to be fun. You will also meet with your group leader and your parents and teacher one time for about half an hour to go over things you learned in the group.

### Will any parts of the study hurt?

Nothing in the study will hurt you. You may feel uncomfortable about answering some of the questions, but your answers may help us learn about how children get along with their parents and with other children.

### Will you get better if you are in this study?

We don't know for sure. You might not get any better. Or, you might do better in school or you might

### Do you have any questions?

You can ask questions any time. You can ask now. You can ask later. You can talk to me or you can talk to someone else.

### Do you have to be in this study?

No, you don't. No one will be mad at you if you don't want to do this. If you don't want to be in this study, just tell us. Or if you do want to be in the study, tell us that. And, remember, you can say yes now and change your mind later. It's up to you.

If you don't want to be in this study, just say so. If you want to be in this study, please tell me "Yes, I want to be in the study."

Assent Form

Your family will be given a copy of this form to keep.

| SIGNATURE OF PERSON CONDUCTING ASSENT DISCUSSION | |
|---|---|
| I have explained the study tounderstand, and the child has verbally agreed to be in the study. | (child name) in language he/she can |
| Signature of Person Conducting Assent Discussion | Date |
| Name of Person Conducting Assent Discussion ( <i>print</i> ) | |



# CONSENT TO PARTICIPATE IN A RESEARCH STUDY

### **Teacher Consent Form**

**Study Title:** Remote School-Home Program to Improve Youth Attention and Behavior in

Mexican Students

**Sponsored by:** National Institute of Health

**Project Directors:** 

Eva Araujo, PhD

Facultad de Psicología

Department of Psychiatry and Behavioral
Sciences

Universidad Autónoma De Sinaloa (UAS)

Ciudad Universitaria,

University of California, San Francisco (UCSF)

401 Parnassus Avenue

Av. de las Américas y Blvd. Universitarios S/N,

Culiacán, Sinaloa, México. C.P. 80080 San Francisco, CA, U.S.A. 94143-0984

**Telephone Number:** 667-798-9385

This is a research study about a remote school-home program to improve Mexican students' attention and behavior. Research studies include only people who choose to take part. Please take your time to make your decision about participating. If you have any questions, you may ask the researchers.

You and your student are being asked to take part in this study because your student is having attentional, behavioral, academic and/or social concerns at school.

### Why is this study being done?

The purpose of this study is to learn about the effectiveness of a of a remote school-home program to improve youth attention and/or behavior for students in Mexico: the CLS-FUERTE program. The program includes a parenting skills component, a teacher consultation component, and a skill building component for children. Knowledge from this study will further research concerning effective interventions and school clinician training programs to improve youth attention and behavior.

### Who pays for the study?

This study is being funded by a federal grant from the National Institute of Health, awarded to Drs. Haack and Araujo.

### How many people will take part in this study?

A total of 88 students, their parents/teachers, and school clinicians across 11 schools will participate in this study.

Caretaker Consent Form 

### What will happen if my child and I take part in this research study?

If you agree to participate, and your child's parent agrees to participate, the following procedures will occur:

1. First, we will conduct screening procedures to find out if you and your student can participate in the program. Your student's family provided your consent for the school and our program staff to share information about your student and for you to complete measures for the program. Screening, which is required for the study, will consist of the following:

- You and your student's parent will answer questions about of your child's behavior.
- If, based on those answers, it seems as though your student meets criteria for our study, you and your student's parent will complete questionnaires about your student's functioning.

If all study criteria are met, your student will be eligible to continue in the study; if study criteria are not met, the student's family will be referred back to your school for other referral options. Information already gathered will be kept by the researchers so that they can report on characteristics of families who consented but did not participate in the study.

- 2. Next, you, your student and your student's parent will participate in the remote program held via videoconferencing, which consists of the following components:
  - A teacher component, which will consist of an up to 60-minute group orientation with the teachers in the program and a 20 to 30-minute meeting with you, the school clinician, a study researcher, the parent and student over a period of about 6 weeks. During these meetings, accommodations in the classroom to improve your student's school performance will be designed and reviewed. A school-home note system for maintaining and rewarding your student's behavior at school will be established.
  - A parent component, which will consist of up to six 90-minute group sessions over a period of about 6 weeks. The sessions will focus on strategies to improve child functioning at home, at school, and with peers and to enhance the quality of family relationships. Parents will be taught strategies for giving instructions, using rewards and consequences, and establishing routines and organizational schemes to help manage their child's behavior. The last group will be a joint child and parent group session to celebrate and encourage the children's participation and successes in the program. All caretakers of any participating child can attend this group session.
  - A child component that consists of up to six 40 to 60-minute group sessions, during
    which time your student will participate in skills training sessions with other students.
    These groups will occur during the school day or after school. They will focus on
    improving social emotional and organizational skills.
- 3. During and after the program, you and your student's parent and school clinician will complete measures about the feasibility and acceptability of the program. After the program, you and student's parent will complete questionnaires about your student's functioning again. We also will invite all participating school clinicians, parents, and teachers to provide feedback about their experiences with the program in focus groups or interviews.

Caretaker Consent Form 

### How will my information be used?

Researchers will use your information to conduct this study. Once the study is done using this information, we may share it with other researchers so they can use it for other studies in the future. We will not share your name or any other personal information that would let the researchers know who you are. We will not ask you for additional permission to share this deidentified information.

### Will any video or audiotaping be done during this study?

All group sessions will be video-recorded using secure video conferencing software (e.g., zoom). These meetings will be digitally recorded and will be stored on secure database servers for supervision, research and training purposes. The digital recordings also may be stored on our secure and password protected Collaborative Life Skills – Remote (CLS-R) training website, using a private video-streaming account in a program such as Vimeo. The recordings will be identified only by numbers, and none of your names will appear on the electronic file labels. The recordings will be kept indefinitely for research, training, and development purposes. The recording is required for trainings, analyses and development of our research.

#### **Study location**

All study procedures will be done remotely or at your school site.

### How long will my student and I be in the study?

Participation in the program involves approximately 90-minutes of meeting time, as well as completion of measures during the program and questionnaires (once before and once after the program), taking approximately 1-2 hours.

#### Can I stop being in the study?

Yes. You can decide to stop at any time. Just tell one of the staff members on the study right away if you wish to stop being in the study.

#### What risks can my child or I expect from being in the study?

The risks in participating in this study as a teacher are minimal; however, you may be uncomfortable answering questions about your student and/or having increased attention paid to your classroom management strategies with the student participating in the program.

### Are there benefits to taking part in the study?

There may be no direct benefits to you or your student from participating in this study. We cannot and do not promise that you or your student will receive any personal benefit from participating in this study. This study will provide a careful monitoring of your student's behavior. Potential benefits include possible reduction in the student's attention and/or behavioral problems, and improvement in academic and social relations as a result of participating in the intervention. You may also receive the educational benefit of participating in a research study and gaining insight into your student through the questionnaire procedure.

Caretaker Consent Form 

#### What other choices do I have if we do not take part in this study?

Your participation in this study is voluntary. You may refuse to participate or may withdraw from the research at any time without consequence.

### Will information about my child and me be kept private?

Participation in research may involve a loss of privacy. We will do our best to make sure that the personal information gathered for this study is kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. Organizations that may look at our research records for quality assurance include the National Institute of Health or the University of California.

Information about you and your student will be kept as confidential as possible. Neither your name nor your student's name will be used in any published reports about this study. All records will be identified by code number only, and the records will be kept on a secure database server. There are some special circumstances that may invoke breaking confidentiality. Such special circumstances consist of our becoming aware of (a) suicidal or homicidal intent or planning on the part of any participant or family member, or (b) child abuse. All members of the research staff will be trained to immediately page or notify the Project Directors upon discovery of either (a) or (b), and to stay in contact with any participant who is in danger until appropriate care can be provided. The Project Directors will evaluate the situation and take the appropriate steps to resolve the risk, including arranging for any emergency care, warning any potential victim, or providing referral to crisis intervention.

### What are the costs of taking part in this study?

There will be no cost to you for any of the research procedures described here.

### Will I be paid for taking part in this study?

You will be paid a \$10 gift card each time you complete assessments (before and after the program), for a total of \$20 in gift cards.

### What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you in any way. Your decision will not affect your employment and/or job benefits.

#### Who can answer my questions about the study?

If you have any questions, comments or concerns about participating in the study, you should first talk with the researchers. You also can contact Dr. Araujo at 667-798-9385. If for some reason you do not wish to do this, or if you still have questions or concerns after talking to Dr. Araujo, you may contact the UAS Ethics Committee, which is concerned with the protection of participants in research projects. You may reach the committee office by calling (667) 712-1656. You may also contact the Ethics Committee if you have questions regarding your rights as a research participant.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Caretaker Consent Form


Web site will include a summary of the results. You can search this Web site at any time.

### **CONSENT**

You will be given a copy of this consent form to keep. The person who signs below has explained this information to you, and your questions were answered.

PARTICIPATION IN RESEARCH IS VOLUNTARY. You have the right to decline to be in this study, or to withdraw from it at any point without penalty or loss of benefits to which you are otherwise entitled.

| If you wish to | participate in this study, please sign below. |
|----------------|-----------------------------------------------|
| Date | Participant's Signature for Consent |
| | Participant's Name (please print) |
| Date | Person Obtaining Consent |

Caretaker Consent Form 

# CONSENT TO PARTICIPATE IN A RESEARCH STUDY

### **School Clinician Consent Form**

**Study Title:** 

Remote School-Home Program to Improve Youth Attention and Behavior in Mexican

Students

**Sponsored by:** National Institute of Health

**Project Directors:** 

Eva Araujo, PhD Lauren Haack, PhD

Facultad de Psicología Department of Psychiatry and Behavioral

Sciences

Universidad Autónoma De Sinaloa (UAS)

University of California, San Francisco (UCSF)

Ciudad Universitaria, 401 Parnassus Avenue

Av. de las Américas y Blvd. Universitarios S/N,

Culiacán, Sinaloa, México. C.P. 80080 San Francisco, CA, U.S.A. 94143-0984

**Telephone Number:** 667-798-9385

This is a research study about a remote school-home program to improve Mexican students' attention and behavior. Research studies include only people who choose to take part. Please take your time to make your decision about participating. If you have any questions, you may ask the researchers.

You are being asked to take part in this study because you are a school clinician.

# Why is this study being done?

The purpose of this study is to learn about the effectiveness of a remote school-home program to improve youth attention and/or behavior for students in Mexico: the CLS-FUERTE program. The program includes a parenting skills component, a teacher consultation component, and a skill building component for children. Knowledge from this study will further research concerning effective interventions and school clinician training programs to improve youth attention and behavior.

# Who pays for the study?

This study is being funded by a federal grant from the National Institute of Health, awarded to Drs. Haack and Araujo.

### How many people will take part in this study?

A total of 88 students, their parents/teachers, and school clinicians across 11 schools will participate in this study.

# What will happen if I take part in this research study?

- You will help identify parents of students from your school site to participate in the remote school-home program to improve youth attention and behavior. Parents of eight students will be recruited at each school. Students will be identified due to concerns about academic and social problems related to inattention and /or hyperactivity-impulsivity. Referrals may come from you, teachers, or through our initial meet-and-greets at your school site. You will approach referred families to explain the project and parents of students who meet first stage entry criteria (e.g., in grade 1-5, mainstream class placement, and absence of significant visual or hearing impairment, severe language delay, psychosis, global intellectual impairment, or serious emotional disturbance requiring special education services per your knowledge and school records, and living with a caretaker who is available to participate in the program, will be invited to participate in screening and will provide verbal consent for exchange of information between the school and our team. Our study staff will contact the parent to complete a remote or in-person screening about academic, social, and behavioral functioning. Parents will also complete a symptom severity rating scale, the Child Symptom Inventory, and the Impairment Rating Scale. To document ADHD symptom presence, we require four or more inattention symptoms and/or four or more hyperactive-impulsive symptoms endorsed by the parent as occurring 'often' or 'very often'. Parents of children not meeting these criteria will be referred back to their school. These recruitment procedures were successfully followed during our previous randomized controlled trial pilot of the in-person version of the CLS-FUERTE program in Mexico. Recruiting students, families and teachers into the program is considered part of your regular work-day.
- Questionnaires in the following categories will be administered and evaluated by school clinicians, parents, and/or teachers: Remote Technology, School Clinician Background and Training Outcomes, Student Background and Outcomes, Program Acceptability and Feasibility.
- School clinicians will receive the program training and will deliver the program remotely
  via videoconferencing with students and their parents and teachers. Our trainers will
  remotely observe the groups modeling and coaching as needed, and conduct individual
  consultation immediately after the sessions. Weekly consultation will also be conducted
  remotely. Fidelity of training measures will be completed by trainers and will be monitored
  by study raters. Satisfaction, usability, and feasibility measures will be completed after
  each session.
- Following the program, questionnaires in the following categories will be administered and
  evaluated again by school clinicians, parents, and/or teachers: School Clinician Training
  Outcomes, Student Outcomes, and Program Acceptability and Feasibility. We also will
  invite all participating school clinicians, parents, and teachers to provide feedback about
  their experiences with the program in focus groups or interviews.

### How will my information be used?

Researchers will use your information to conduct this study. Once the study is done using this information, we may share it with other researchers so they can use it for other studies in the future. We will not share your name or any other personal information that would let the researchers know who you are. We will not ask you for additional permission to share this de-identified information.

# Will any video or audiotaping be done during this study?

All group sessions will be video-recorded using secure video conferencing software (e.g., zoom). These meetings will be digitally recorded and will be stored on secure database servers for supervision, research and training purposes. The digital recordings may be stored on our secure and password protected Collaborative Life Skills – Remote (CLS-R) training website, using a private video-streaming account in a program such as Vimeo. The recordings will be identified only by numbers, and none of your names will appear on the electronic file labels. The recordings will be kept indefinitely for research, training, and development purposes The recording is required for trainings, analyses and development of our research.

# How long will I be in the study?

Participation in the study will take a total of about 33 hours to be trained and to implement the program over about 6 weeks, and a total of about 2 hours for completing questionnaires over the course of the study.

# Can I stop being in the study?

You are being asked to participate in this study by providing information about your background and training experience as part of this study. **Your participation is entirely voluntary.** You may refuse to take part in the study or you may stop your participation in the study at any time.

### What side effects or risks can I expect from being in the study?

The risks in participating in this study as a school clinician are minimal; however, you may be uncomfortable answering questions about your training background and/or being observed while implementing the program.

### Are there benefits to taking part in the study?

There may be no direct benefits to you from participating in this study. Potential benefits include learning about evidence-based strategies helpful for improving student's attention and/or behavior. Your students may exhibit possible reduction in attention and/or behavioral problems, and improvement in academic and social relations as a result of participating in the intervention. You may also receive the educational benefit of participating in a research study. Your students and others may benefit in the future from this research.

# What other choices do I have if I do not take part in this study?

Your participation in this study is voluntary. You may refuse to participate or may withdraw from the research at any time without consequence.

### Will information about me and my responses about my student be kept private?

Participation in research may involve a loss of privacy. Information about you and information

which you provide about your students will be kept as confidential as possible. However, we cannot guarantee total privacy. Neither your name nor your students' names will be used in any published reports about this study. All records will be identified by code number only, and the records will be kept on a secure network platform. The University of California and the study sponsor, the National Institute of Health, will have access to the research records for auditing or monitoring purposes. There are some special circumstances that may invoke breaking confidentiality. Such special circumstances consist of our becoming aware of (a) suicidal or homicidal intent or planning on the part of any participant or family member, or (b) child abuse. All members of the research staff will be trained to immediately page or notify the Project Directors upon discovery of either (a) or (b), and to remain in contact with any participant who is in danger until appropriate care can be provided. The Project Directors will evaluate the situation and take the appropriate steps to resolve the risk, including arranging for any emergency care, warning any potential victim, or providing referral to crisis intervention.

# What are the costs of taking part in this study?

You will not be charged for any of the study procedures.

### Will I be paid for taking part in this study?

You will be paid \$10 in gift cards each time you complete questionnaires (before and after the program), for a total of \$20 in gift cards.

# What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you in any way. Your decision will not affect your employment and/or job benefits.

### Who can answer my questions about the study?

If you have any questions, comments or concerns about participating in the study, you should first talk with the researchers. You also can contact Dr. Araujo at 667-798-9385. If for some reason you do not wish to do this, or if you still have questions or concerns after talking to Dr. Araujo, you may contact the UAS Ethics Committee, which is concerned with the protection of participants in research projects. You may reach the committee office by calling 667-712-1656. You may also contact the Ethics Committee if you have questions regarding your rights as a research participant.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### **CONSENT**

You will be given a copy of this consent form to keep. The person who signs below has

explained this information to you, and your questions were answered.

PARTICIPATION IN RESEARCH IS VOLUNTARY. You or your students have the right to decline to be in this study, or to withdraw from it at any point without penalty or loss of benefits to which you are otherwise entitled.

| If you wish to participate and have your students participate in this study, please sign below. | |
|---|---|
| Signature of School Clinician | Date |
| School Clinician Name (Print) | |
| School | |
| Person Obtaining Consent | <br>Date |



# CONSENT TO PARTICIPATE IN A RESEARCH STUDY

# **Parent/Caregiver Consent Form**

**Study Title:** Remote School-Home Program to Improve Youth Attention and Behavior in

Mexican Students

**Sponsored by:** National Institute of Health

**Project Directors:** 

Eva Araujo, PhD Lauren Haack, PhD
Facultad de Psicología Department of Psychiatry and Behavioral
Sciences

Universidad Autónoma De Sinaloa (UAS)

Ciudad Universitaria,

University of California, San Francisco (UCSF)

401 Parnassus Avenue

Av. de las Américas y Blvd. Universitarios S/N,

Culiacán, Sinaloa, México. C.P. 80080 San Francisco, CA, U.S.A. 94143-0984

**Telephone Number:** 667-798-9385

This is a research study about a remote school-home program to improve Mexican students' attention and behavior. Research studies include only people who choose to take part. Please take your time to make your decision about participating, and discuss your decision with your family, friends, mental health care professional, or physician if you wish. If you have any questions, you may ask the researchers.

You and your child are being asked to take part in this study because your child is having attentional, behavioral, academic and/or social concerns at school.

### Why is this study being done?

The purpose of this study is to learn about the effectiveness of a of a remote school-home program to improve youth attention and/or behavior for students in Mexico: the CLS-FUERTE program. The program includes a parenting skills component, a teacher consultation component, and a skill building component for children. Knowledge from this study will further research concerning effective interventions and school clinician training programs to improve youth attention and behavior.

#### Who pays for the study?

This study is being funded by a federal grant from the National Institute of Health, awarded to Drs. Haack and Araujo.

### How many people will take part in this study?

A total of 88 students, their parents/teachers, and school clinicians across 11 schools will participate in this study.

Caretaker Consent Form 

### What will happen if my child and I take part in this research study?

If you agree to participate, and your child's teacher agrees to participate, the following procedures will occur:

- 1. First, we will conduct screening procedures to find out if you and your child can participate in the program. You provided your consent for your school and our program staff to share information about your child and for your child's teacher to complete measures for the program. Screening, which is required for the study, will consist of the following:
  - You and your child's teacher will answer questions about of your child's behavior.
  - If, based on those answers, it seems as though your child meets criteria for our study, you and your child's teacher will complete questionnaires about your child's functioning.

If all study criteria are met, your child will be eligible to continue in the study; if study criteria are not met, you will be referred back to your school for other referral options. Information already gathered will be kept by the researchers so that they can report on characteristics of families who consented but did not participate in the study.

- 2. Next, you, your child and your child's teacher will participate in the remote program held via videoconferencing, which consists of the following components:
  - A teacher component, which will consist of an up to 60-minute group orientation with the teachers and a 20 to 30-minute meeting with the teacher, school clinician, study researcher, parent and child over a period of about 6 weeks. During these meetings, accommodations in the classroom to improve your child's school performance will be designed and reviewed. A school-home note system for maintaining and rewarding your child's behavior at school will be established.
  - A parent component, which will consist of up to six 90-minute group sessions with other parents over a period of about 6 weeks. The sessions will focus on strategies to improve child functioning at home, at school, and with peers and to enhance the quality of family relationships. Parents will be taught strategies for giving instructions, using rewards and consequences, and establishing routines and organizational schemes to help manage their child's behavior. The last group will be a joint child and parent group session to celebrate and encourage the children's participation and successes in the program. All caretakers of any participating child can attend this group session.
  - A child component that consists of up to six 40 to 60-minute group sessions, during which time your child will participate in skills training sessions with other children. These groups will occur during the school day or after school. They will focus on improving social emotional and organizational skills.
- 3. During and after the program, you and your child's teacher and school clinician will complete measures about the feasibility and acceptability of the program. After the program, you and your child's teacher will complete questionnaires about your child's functioning again. We also will invite all participating school clinicians, parents, and teachers to provide feedback about their experiences with the program in focus groups or interviews.

Caretaker Consent Form 

### How will my and my child's information be used?

Researchers will use your and your child's information to conduct this study. Once the study is done using this information, we may share it with other researchers so they can use it for other studies in the future. We will not share your names or any other personal information that would let the researchers know who you are. We will not ask you for additional permission to share this de-identified information.

#### Will any video or audiotaping be done during this study?

All group sessions will be video-recorded using secure video conferencing software (e.g., zoom). These meetings will be digitally recorded and will be stored on secure database servers for supervision, research and training purposes. The digital recordings also may be stored on our secure and password protected Collaborative Life Skills – Remote (CLS-R) training website, using a private video-streaming account in a program such as Vimeo. The recordings will be identified only by numbers, and none of your names will appear on the electronic file labels. The recordings will be kept indefinitely for research, training, and development purposes. The recording is required for trainings, analyses and development of our research.

### What if my child is taking medication for ADHD?

If your child is taking medication, he or she still is eligible for the current project as long as he or she has been taking the same type or dose of medication for the past month (immediately prior to the screening). Your child can continue to take his/her medication as usual throughout his/her participation in the current project.

### **Study location**

All study procedures will be done remotely or at your child's school.

### How long will my child and I be in the study?

The total time commitment for all participating families includes completion of measures during the program and questionnaires (once before and once after the program), taking approximately 1-2 hours. Participation in the program involves attending six weekly 90-minute group meetings for parents, six weekly 40-60 minute group meetings for children, and one 20-30 minute meeting between parents, teachers, school clinicians and children.

### Can my child or I stop being in the study?

Yes. You, or your child, can decide to stop at any time. Just tell one of the staff members on the study right away if you wish to stop being in the study.

Also, the study researcher may stop you or your child from taking part in this study at any time if he or she believes it is in your best interest, if you do not follow the study rules, or if the study is stopped.

### What risks can my child or I expect from being in the study?

Potential Risks for Completing Questionnaires: Potential risks include discomfort that some people may feel when being interviewed, observed, or when completing questionnaires about personal matters. Protection against these risks includes highly-trained staff, including child Caretaker Consent Form


psychologists. The questionnaires and program will be conducted by experienced mental health professionals who are trained to be sensitive to the feelings and well-being of the participants.

- Potential Risks for Remote Groups: As part of participation in this program, families will be exposed to remote groups which involve parents and children interacting with and sharing personal information with other families having similar problems. This may be embarrassing or stigmatizing for some families. However, feedback from participants taking part in previous similar studies to this has been positive. All participating parents and children will be instructed about privacy and requested that they only join groups while in a private setting, not reveal the identity of any other group members or repeat any personal information provided by other group members during group meetings. Protection against these risks also includes use of highly trained staff and availability of child psychologists; all staff will be trained in protecting the confidentiality of patient information.
- Potential Risks for Video-recordings: Potential risks include discomfort that some people may feel when being recorded. Loss of confidentiality is the major risk if your or your child's identity accidentally is discovered by anyone viewing the recordings. Video-recordings made during the parent, teacher and child sessions will be used solely for research and training purposes, and will be kept on a secure server. Video-recordings will be electronically labeled with code numbers only; labels will not include names.
- For more information about risks, please ask one of the researchers.

### Are there benefits to taking part in the study?

There may be no direct benefits to you or your child from participating in this study. We cannot and do not promise that you or your child will receive any personal benefit from participating in this study. This study will provide a careful monitoring of your child's behavior. Potential benefits include possible reduction in attention and/or behavioral problems, and improvement in academic and social relations as a result of participating in the intervention. You may also receive the educational benefit of participating in a research study and gaining insight into your child through the questionnaire procedure.

### What other choices do I have if we do not take part in this study?

Your other choices may include not taking part in this research study, getting standard intervention for attention and/or behavioral problems (at school or outside of school) without being in a study, or taking part in another study. If you decide not to take part in this study, there will be no penalty to you. Your choice will not affect your or your child's care or how you are treated at school.

### Will information about my child and me be kept private?

Participation in research may involve a loss of privacy. We will do our best to make sure that the personal information gathered for this study is kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. Organizations that may look at our research records for quality assurance include the National Institute of Health or the University of California.

Information about you and your child will be kept as confidential as possible. Neither your name nor your child's name will be used in any published reports about this study. All records will be identified by code number only, and the records will be kept on a secure database server. There are Caretaker Consent Form


some special circumstances that may invoke breaking confidentiality. Such special circumstances consist of our becoming aware of (a) suicidal or homicidal intent or planning on the part of any participant or family member, or (b) child abuse. All members of the research staff will be trained to immediately page or notify the Project Directors upon discovery of either (a) or (b), and to stay in contact with any participant who is in danger until appropriate care can be provided. The Project Directors will evaluate the situation and take the appropriate steps to resolve the risk, including arranging for any emergency care, warning any potential victim, or providing referral to crisis intervention.

### What are the costs of taking part in this study?

There will be no cost to you or to your insurance carrier(s) for any of the research procedures described here.

### Will I be paid for taking part in this study?

You will be paid with a \$10 gift card each time you complete assessments (before and after the program), for a total of \$20 in gift cards.

### Who can answer my questions about the study?

If you have any questions, comments or concerns about participating in the study, you should first talk with the researchers. You also can contact Dr. Araujo at 667-798-9385. If for some reason you do not wish to do this, or if you still have questions or concerns after talking to Dr. Araujo, you may contact the UAS Ethics Committee, which is concerned with the protection of participants in research projects. You may reach the committee office by calling (667) 712-1656. You may also contact the Ethics Committee if you have questions regarding your rights as a research participant.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### **CONSENT**

You will be given a copy of this consent form to keep. The person who signs below has explained this information to you, and your questions were answered.

PARTICIPATION IN RESEARCH IS VOLUNTARY. You or your child have the right to decline to be in this study, or to withdraw from it at any point without penalty or loss of benefits to which you are otherwise entitled.

| Date | Participant's Signature for Consent |
|------|-------------------------------------|
| | Participant's Name (please print) |
| te | Person Obtaining Consent |

If you wish to participate and have your child participate in this study, please sign below.

AND By signing below, you are giving your permission for your child to be included in this study. Your

Caretaker Consent Form 

| permission is needed as your child is unable to consent for himself/herself because he/she is a minor: | |
|---|---|
| Date | Parent or Legal Guardian |

Caretaker Consent Form 

# CONSENTIMIENTO PARA PARTICIPACIÓN EN EL ESTUDIO

# Formato de Consentimiento de personal clínico escolar

**Título del estudio:** Programa Escuela-Hogar en línea para mejorar la atención y la conducta de estudiantes

mexicanos

Financiado por: Instituto Nacional de Salud

### Director del proyecto:

Eva Araujo, PhD

Facultad de Psicología Universidad Autónoma De Sinaloa (UAS) Ciudad Universitaria, Av. de las Américas y Blvd. Universitarios S/N, Culiacán, Sinaloa, México. C.P. 80080

**Telephone Number:** 667-798-9385

Lauren Haack, PhD
Department of Psychiatry and Behavioral Sciences
University of California, San Francisco (UCSF) 401
Parnassus Avenue

San Francisco, CA, U.S.A. 94143-0984

Este es un estudio de investigación sobre un programa entre la escuela y el hogar en línea, para mejorar la atención y la conducta de estudiantes mexicanos. Los estudios de investigación incluyen solo a personas que desean ser parte de ellos. Le pedimos, que por favor se tome su tiempo para decidir si participará. Si tiene alguna pregunta no dude en preguntarle a las investigadoras.

Si está siendo invitado a participar en este estudio es porque forma parte del personal considerado clínico escolar.

# ¿Porqué se está realizando este estudio?

El propósito de este estudio es aprender acerca de la eficacia de un programa entre escuela y hogar en línea para mejorar la atención y la conducta de estudiantes en México: CLS-FUERTE. El programa incluye un componente de habilidades parentales, un componente de orientación a los profesores de aula, y un componente de construcción de habilidades de los niños. Los resultados que surjan de este estudio promoverán más investigaciones de intervenciones efectivas y el entrenamiento de personal escolar para mejorar la atención y la conducta de los niños/as.

# ¿Quién paga el estudio?

Este estudio está financiado por una beca federal del Instituto Nacional de Salud, ganado por las Dras. Lauren Haack y Eva Araujo.

# ¿Cuántas personas formarán parte del estudio?

Un total de 88 estudiantes, sus padres/familiares, y personal clínico escolar de 11 escuelas participarán en este estudio

# ¿Qué pasará si formo parte del estudio?

Usted ayudará a identificar a padres de niños de su escuela que pudieran participar en el programa Escuela-Hogar en línea para mejorar la atención y la conducta. Se reclutarán a los padres de ocho estudiantes en cada escuela. Los estudiantes los identificará a partir de los problemas académicos y sociales que puedan presentar relacionados con inatención y/o hiperactividad/impulsividad. Las referencias deberán venir de usted, de los profesores, o a través de nuestra reunión inicial en la escuela. Usted se acercará a las familias derivadas y a los padres de estudiantes que cumplen con los criterios de ingreso para la primera etapa para explicarles el proyecto (e.g. que esté en 1-5 grado, que asista a clases ordinarias, y con ausencia de discapacidad visual o auditiva significativa, retraso grave del lenguaje, psicosis, discapacidad intelectual global o trastorno emocional que requiera servicios de educación especial según su conocimiento y registros escolares, y viviendo con un cuidador que esté disponible para participar en el programa, será invitado a participar en la selección y dará consentimiento verbal para el intercambio de información entre la escuela y nuestro equipo). El staff del estudio se pondrá en contacto con los padres para completar en línea o personalmente los instrumentos acerca del funcionamiento académico, social y conductual de su hijo/a. Los padres también llenarán una escala de severidad d síntomas, el Inventario de Síntomas Infantiles (CSI), y la escala Impairment Rating Scale. Para documentar la presencia de síntomas de Déficit de Atención e Hiperactividad/impulsividad, necesitamos cuatro o más síntomas de inatención y cuatro o más síntomas de hiperactividad/impulsividad, que los padres detectarán como "a menudo" o "muy a menudo". Los padres de los niños que no cumplan con este criterio será referido nuevamente a su escuela. Este procedimiento de reclutamiento fue exitosamente seguido durante nuestro anterior estudio piloto aleatorio controlado en la versión presencial del programa CLS-FUERTE en México. El reclutamiento de estudiantes, familias, y maestros en el programa es considerado parte del trabajo regular del día a día.

El personal clínico escolar, los padres, y/o los profesores completarán los cuestionarios de las siguientes categorías: tecnología en línea, retroalimentación y resultados de la capacitación al personal clínico escolar, retroalimentación y resultados de estudiantes, aceptabilidad y viabilidad del programa.

El personal clínico escolar recibirá la capacitación del programa y lo impartirá de forma remota (en línea) a través de videoconferencias con los estudiantes, sus padres y maestros. Nuestros instructores (equipo de investigación) observarán de forma remota (en línea) cómo se llevan a cabo las sesiones grupales, y se realizarán orientaciones individuales inmediatamente después de las sesiones. La orientación semanal también se realizará en línea. Los instructores completarán la fidelidad de las medidas de capacitación y serán supervisadas por los evaluadores del estudio. Las medidas de satisfacción, uso, y viabilidad se completarán después de cada sesión.

Después del programa, el personal clínico escolar, los padres y/o maestros completarán nuevamente los cuestionarios de las siguientes categorías: Resultados de la capacitación del personal clínico escolar, Resultados de los estudiantes, y aceptabilidad y viabilidad del programa. También invitaremos a todos los participantes, personal clínico escolar, padres, y maestros a brindarnos comentarios sobre sus experiencias con el programa en grupos focales o entrevistas.

# ¿Se realizarán video y audio grabaciones durante el estudio?

Todas las sesiones de grupo serán video-grabadas usando una plataforma de videoconferencia segura (e.g. zoom). Estas sesiones serán grabadas digitalmente y estarán resguardadas en un servidor de base de datos seguro para ser revisados después por los clínicos/investigadores, con el fin de evaluar las reuniones y para propósitos de investigación y entrenamiento. Las grabaciones serán resguardas en nuestro sistema protegido con contraseña en la página web del entrenamiento del programa Colaborativo para Habilidades de la Vida en línea (CLS-Remote), usando una cuenta privada de video-streaming en un programa como Vimeo. Las grabaciones serán identificadas solo con números, y ninguno de sus nombres aparecerán en ellas. Las grabaciones serán guardadas indefinidamente para propósitos de investigación y entrenamiento, y desarrollo de los objetivos. La grabación es necesaria para entrenamientos, análisis y desarrollo de la

# ¿Cuánto tiempo estaré en el estudio?

La participación en el estudio le tomará alrededor 33 horas que contemplan el entrenamiento y la implementación del programa en 6 semanas, y un total de dos horas para completar los cuestionarios en todo el curso del estudio.

# ¿Puedo dejar de participar en el estudio?

Usted está siendo invitado a participar en el estudio para que proporcione información acerca de su experiencia y su entrenamiento como parte de este estudio. **Su participación es complemente voluntaria**. Usted puede negarse a formar parte del estudio o detener su participación en cualquier momento del estudio.

# ¿Qué riesgos puedo tener al fomar parte del estudio?

Los riesgos que puede tener al formar parte de estudio son mínimos; sin embargo, podría sentirse incómodo de responder algunas preguntar sobre su experiencia en el entrenamiento y/o sentirse observado durante la implementación del programa.

# ¿Hay algún beneficio por formar parte del estudio?

No hay beneficios directos por participar en el estudio. Los beneficios posibles incluyen aprender nuevas estrategias basadas en evidencia científica sobre ayudar a la mejora de la atención y conducta de los estudiantes. Puede ser que su estudiante reduzca los problemas de atención y/o de conducta, y que mejore en los académico y las relaciones sociales como resultado de su participación en la intervención. También puede ser que usted reciba el beneficio educativo de participar en un estudio. Su estudiante y otros podrán verse beneficiados por esta investigación en un futuro.

# ¿Qué otras opciones tengo si no quiero formar parte del estudio?

Su participación en el estudio es voluntaria. Usted puede negarse a participar o dejar la investigación sin consecuencia alguna.

# ¿Qué información sobre mi persona y sobre mi estudiante se mantendrá en privado?

La participación en investigaciones puede llevar a la pérdida de la privacidad, pero la información acerca de usted y su estudiante se mantendrá como confidencial lo más posible. Sin embargo, no podemos garantizar total privacidad. Ni su nombre ni el de su estudiante serán usados en algún reporte de publicación acerca de este estudio. Todos los registros se identificarán sólo con un código numérico, y los registros permanecerán guardados en una plataforma web segura.

La Universidad de California, y el financiador del estudio, el Instituto Nacional de Salud Mental, tendrán acceso a los registros de investigación para propósitos de auditoría o de monitorización. Hay algunas circunstancias especiales que pueden provocar quebrantar la confidencialidad. Esas circunstancias consisten en (a) suicidio, o intento o plan de homicidio de alguno de los miembros de la familia, o (b) abuso del niño. Todos los miembros del grupo de investigación están entrenados para registrar o notificar de manera inmediata al Investigador Principal (PI) si descubre alguna de esas circunstancias (a) o (b), estar junto a cualquiera de los participantes si éste se encuentra en peligro hasta que tenga un cuidado apropiado. El PI evaluará la situación y realizará los pasos necesarios para resolver el riesgo, incluyendo dar atención de emergencia, advertir de cualquier víctima potencial, dando intervención en crisis, o

referenciando a intervención en crisis.

# ¿Cuál es el costo al formar parte del estudio?

No se le cobrará por ninguno de los procedimientos del estudio.

# ¿Me pagarán por ser parte del estudio?

Se le pagarán \$200.00 pesos cada vez que complete los cuestionarios (antes y después del programa), siendo un total de \$400.00 pesos.

### ¿Cuáles son mis derechos si formo parte del estudio?

Es su decisión formar parte de este estudio. Usted decidirá si forma parte del estudio o no. Si decide formar parte del estudio, puede dejarlo en el momento que lo desee. No importa qué decisión haya tomado, no habrá alguna amonestación.

# ¿Quién puede responder mis dudas sobre el estudio?

Si usted tiene alguna pregunta, comentario o preocupación sobre su participación en el estudio, debería hablar con los investigadores. Puede contactar a la Dra. Araujo al número (667) 798-93-85. Si por alguna razón usted no desea hacer esto, o si sigue teniendo dudas o preocupaciones después de hablar con la Dra. Araujo, puede contactar al Comité de Ética de la Universidad Autónoma de Sinaloa, quienes se encargan de la protección de los voluntarios en los proyectos de investigación. También puede contactar a este comité en caso de tener dudas sobre sus derechos como participante de una investigación.

Puede encontrar en el siguiente link: <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> una descripción del programa, tal como es solicitado por las leyes de Estados Unidos. Esta página de internet no incluye información de su identificación personal. Sin embargo, dicha página si incluirá un resumen de los resultados de este estudio. Puede usted acceder a esta página cuando lo desee.

### **CONSENTIMIENTO**

Usted tendrá una copia de este consentimiento para que la tenga consigo. La persona que firma a continuación es quien le ha explicado toda esta información y respondido a sus preguntas.

LA PARTICIPACIÓN EN LA INVESTIGACIÓN ES VOLUNTARIA. Usted y/o su estudiante tienen el derecho de negar ser parte del estudio, o retirarse en cualquier momento sin alguna multa o pérdida de beneficios a los que tiene derecho.

| Si usted desea participar y tiene estudiantes participando en este estudio, por favor firme debajo. | |
|---|---|
| Firma del personal clínico escolar | Fecha |
| Nombre del personal clínico escolar (impresa) | |
| Escuela | |
| Persona que obtiene el consentimiento | Fecha |

# CONSENTIMIENTO PARA PARTICIPACIÓN EN EL ESTUDIO

### Formato de Consentimiento de maestros

**Título del estudio:** Programa Escuela-Hogar en línea para mejorar la atención y la conducta de estudiantes

mexicanos

**Financiado por:** Instituto Nacional de Salud

### Director del proyecto:

Eva Araujo, PhD

Facultad de Psicología Universidad Autónoma De Sinaloa (UAS) Ciudad Universitaria, Av. de las Américas y Blvd. Universitarios S/N, Culiacán, Sinaloa, México. C.P. 80080

**Telephone Number:** 667-798-9385

Lauren Haack, PhD
Department of Psychiatry and Behavioral Sciences
University of California, San Francisco (UCSF) 401
Parnassus Avenue

San Francisco, CA, U.S.A. 94143-0984

Este es un estudio de investigación sobre un programa entre la escuela y el hogar en línea, para mejorar la atención y la conducta de estudiantes mexicanos. Los estudios de investigación incluyen solo a personas que desean ser parte de ellos. Le pedimos, que por favor se tome su tiempo para decidir si participará. Si tiene alguna pregunta no dude en preguntarle a las investigadoras.

Si está siendo invitado a participar en este estudio es porque un estudiante está teniendo problemas de atención, conducta, académicos y/o sociales en la escuela.

### ¿Porqué se está realizando este estudio?

El propósito de este estudio es aprender acerca de la eficacia de un programa entre escuela y hogar en línea para mejorar la atención y la conducta de estudiantes en México: CLS-FUERTE. El programa incluye un componente de habilidades parentales, un componente de orientación a los profesores de aula, y un componente de construcción de habilidades de los niños. Los resultados que surjan de este estudio promoverán más investigaciones de intervenciones efectivas y el entrenamiento de personal escolar para mejorar la atención y la conducta de los niños/as.

# ¿Quién paga el estudio?

Este estudio está financiado por una beca federal del Instituto Nacional de Salud, ganado por las Dras. Lauren Haack y Eva Araujo.

# ¿Cuántas personas formarán parte del estudio?

Un total de 88 estudiantes, sus padres/familiares, y personal clínico escolar de 11 escuelas participarán en este estudio

# ¿Qué pasará si formo parte del estudio?

1. Primero, realizaremos un procedimiento de selección para conocer si usted y su estudiante pueden formar parte del programa. La familia de su estudiante otorgó el consentimiento a la escuela y a nuestro staff del programa para compartir la información acerca de su estudiante y a ustede para completar los instrumentos del programa.

La selección que es requerida para el estudio, consiste en lo siguiente:

- Usted y el padre de su estudiante responderán los cuestionarios sobre la conducta del niño.
- Si, basándonos en estos cuestionarios, su estudiante cumple con los criterios del estudio, usted y el padre del estudiante responderán cuestionarios acerca del funcionamiento de su niño.

Si todos los criterios se cumplen, su estudiante será elegido para continuar en el estudio; si los criterios no se cumplen se le pedirá a la escuela que le ofrezca otro tipo de opciones de ayuda. La información que hasta el momento se ha recabado por los investigadores, se quedará con ellos, para que sean reportadas las características de las familias que no participaron en este estudio.

- 2. Después, usted, su estudiante y los padres del niño participarán en un programa en línea (remoto) vía videoconferencia, que consiste en los siguientes componentes:
  - O Un componente de maestros, el cual consiste en una orientación grupal de maestros de 60 minutos y dos reuniones de seguimiento de 20-30 minutos con los maestros, el personal clínico escolar, los padres y los niños en un periodo de 6 semanas. Durante estas reuniones, diseñaremos y revisaremos adaptaciones en la clase de su niño para su mejora. Un sistema de anotaciones entre escuela-hogar llevaremos a cabo para mantener y premiar la conducta de su hijo.
  - O Un componente de padres, el cual consiste en seis sesiones grupales de 90 minutos con los padres en un periodo de 6 semanas. Estas sesiones se enfocaran en estrategias que ayudarán a su hijo a funcionar mejor en la casa, escuela, y con sus pares, así como a mejorar la calidad de la relación familiar. Los padres aplicarán estrategias dando instrucción, usando premios y consecuencias, y estableciendo rutinas y esquemas de organización para ayudar al manejo de la conducta de su hijo. En el último grupo se realizará una sesión con los niños y los padres para celebrar y alentar la participación de los niños y su éxito en el programa. Todos los cuidadores de cualquiera de los niños que participan podrán asistir a la sesión de grupo.
  - O Un componente de niños que consiste en seis sesiones de 40 a 60 minutos, durante ese tiempo su hijo participará en sesiones de entrenamiento de habilidades con otros niños. Estos grupos serán durante los horarios de clase o justo después de clases..
- 3. Usted, los padres del estudiante y el personal clínico escolar, completarán instrumentos sobre fiabilidad y aceptación del programa, se responderán durante y después del programa. Además, después del programa, usted y los padres del estudiante responderán de nuevo los cuestionarios acerca del funcionamiento del niño. También invitaremos a todos los participantes a otorgar retroalimentación acerca de su experiencia con el programa en grupos focales y entrevistas.

# ¿Se realizarán video y audio grabaciones durante el estudio?

Todas las sesiones de grupo serán video-grabadas usando una plataforma de videoconferencia segura (e.g. zoom). Estas sesiones serán grabadas digitalmente y estarán resguardadas en un servidor de base de datos seguro para ser revisados después por los clínicos/investigadores, con el fin de evaluar las reuniones y para propósitos de investigación y entrenamiento. Las grabaciones serán resguardas en nuestro sistema protegido con contraseña en la página web del entrenamiento del programa Colaborativo para Habilidades de la Vida en línea (CLS-Remote), usando una cuenta privada de video-streaming en un programa como Vimeo. Las grabaciones serán identificadas solo con números, y ninguno de sus nombres aparecerán en ellas. Las grabaciones serán guardadas indefinidamente para propósitos de investigación y entrenamiento,

Caretaker Consent Form 

y desarrollo de los objetivos. La grabación es necesaria para entrenamientos, analisis y desarrollo de la investigación.

### Lugar del estudio

Todos los procedimientos del estudio se llevarán a cabo en línea o en la escuela de su hijo.

# ¿Cuánto tiempo estaré en el estudio?

La participación en el estudio le tomará alrededor 90 minutos en una reunión, así como completar instrumentos durante el programa (uno antes y otro después del programa) que le tomará aproximadamente 1-2 horas.

# ¿Puedo dejar de participar en el estudio?

Si. Usted puede decidir no participar en cualquier momento. Solo dígaselo a algún miembro del equipo del estudio cuando lo desee.

# ¿Qué riesgos puedo tener al fomar parte del estudio?

Los riesgos que puede tener al formar parte de estudio como maestro son mínimos; sin embargo, podría sentirse incómodo de responder algunas preguntar sobre su estudiante y/o poniendo mayor atención en el desarrollo del niño en el aula, así como manejando las estrategias con el estudiante participante en el programa.

# ¿Hay algún beneficio por formar parte del estudio?

Puede no haber beneficios directos para usted o su estudiante al participar en el estudio. No podemos prometer que su estudiante recibirá algún beneficio personal de la participación de este estudio. Este estudio dará un seguimiento cuidadoso de la conducta de su estudiante. Los beneficios principales que pueden derivarse pueden ser la reducción de los problemas de atención y/o conducta de su estudiante, y una mejora en lo académico y sus relaciones sociales como resultado de la participación en la intervención. También tendrá el beneficio educativo de participar en un experimento científico y saber más acerca de su estudiante a partir de la evaluación.

# ¿Qué otras opciones tengo si no quiero formar parte del estudio?

Su participación en el estudio es voluntaria. Usted puede negarse a participar o dejar la investigación sin consecuencia alguna.

# ¿Qué información sobre mi persona y sobre mi estudiante se mantendrá en privado?

La participación en investigaciones incluye perder privacidad. Haremos todo lo posible por asegurarnos de que la información personal adquirida en este estudio permanezca en privado. Sin embargo, no podemos garantizar total privacidad. Su información personal puede ser usada si es requerida por la ley. Algunas organizaciones revisan nuestros registros de investigación para que la calidad esté garantizada incluyendo el Instituto Nacional de Salud o el Comité de Recursos Humanos de UCSF.

La información acerca de usted y su estudiante se mantendrá como confidencial lo más posible. Ni su

Caretaker Consent Form 

nombre ni el de su estudiante será usado en algún reporte de publicación acerca de este estudio. Todos los registros se identificarán sólo con un código numérico, y los registros permanecerán guardados en servidor de base de datos seguro. Hay algunas circunstancias especiales que pueden provocar quebrantar la confidencialidad. Esas circunstancias consisten en (a) suicidio, o intento o plan de homicidio de alguno de los miembros de la familia, o (b) abuso del niño. Todos los miembros del grupo de investigación está entrenado para registrar o notificar de manera inmediata al Investigador Principal (PI) si descubre alguna de esas circunstancias (a) o (b), estar junto a cualquiera de los participantes si este se encuentra en peligro hasta que tenga un cuidado apropiado. El PI evaluará la situación y realizará los pasos necesarios para resolver el riesgo, incluyendo dar atención de emergencia, advertir de cualquier víctima potencial, dando intervención en crisis, o haciendo un reporte de abuso a los servicios de protección infantil.

# ¿Cuál es el costo al formar parte del estudio?

No se le cobrará por ninguno de los procedimientos del estudio.

# ¿Me pagarán por ser parte del estudio?

Se le pagarán \$200.00 pesos cada vez que complete los cuestionarios (antes y después del programa), siendo un total de \$400.00 pesos.

# ¿Quién puede responder mis dudas sobre el estudio?

Si usted tiene alguna pregunta, comentario o preocupación sobre su participación en el estudio, debería hablar con los investigadores. Puede contactar a la Dra. Araujo al número (667) 798-93-85. Si por alguna razón usted no desea hacer esto, o si sigue teniendo dudas o preocupaciones después de hablar con la Dra. Araujo, puede contactar al Comité de Ética de la Universidad Autónoma de Sinaloa, quienes se encargan de la protección de los voluntarios en los proyectos de investigación. También puede contactar a este comité en caso de tener dudas sobre sus derechos como participante de una investigación.

Puede encontrar en el siguiente link: <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> una descripción del programa, tal como es solicitado por las leyes de Estados Unidos. Esta página de internet no incluye información de su identificación personal. Sin embargo, dicha página si incluirá un resumen de los resultados de este estudio. Puede usted acceder a esta página cuando lo desee.

#### **CONSENTIMIENTO**

Usted tendrá una copia de este consentimiento para que la tenga consigo. La persona que firma a continuación es quien le ha explicado toda esta información y respondido a sus preguntas.

LA PARTICIPACIÓN EN LA INVESTIGACIÓN ES VOLUNTARIA. Usted y/o su estudiante tienen el derecho de negar ser parte del estudio, o retirarse en cualquier momento sin alguna multa o pérdida de beneficios a los que tiene derecho.

| Si usted desea pa | articipar y tiene un estudiante que participa en este estudio, por favor firme debajo. |
|---|---|
| Fecha | Firma del participante para consentimiento |
| | Nombre del participante(impreso) |

Caretaker Consent Form 

| Fecha | Persona que obtiene el consentimiento |
|-------|---------------------------------------|

Caretaker Consent Form 

# CONSENTIMIENTO PARA PARTICIPACIÓN EN EL ESTUDIO

### Formato de consentimiento para cuidadores

**Título del estudio:** Programa Escuela-Hogar en línea para mejorar la atención y la conducta de estudiantes

mexicanos

Financiado por: Instituto Nacional de Salud

### Director del proyecto:

Eva Araujo, PhD

Facultad de Psicología Universidad Autónoma De Sinaloa (UAS) Ciudad Universitaria, Av. de las Américas y Blvd. Universitarios S/N, Culiacán, Sinaloa, México. C.P. 80080

**Telephone Number:** 667-798-9385

Lauren Haack, PhD
Department of Psychiatry and Behavioral Sciences
University of California, San Francisco (UCSF) 401
Parnassus Avenue

San Francisco, CA, U.S.A. 94143-0984

Este es un estudio de investigación sobre un programa entre la escuela y el hogar en línea, para mejorar la atención y la conducta de estudiantes mexicanos. Los estudios de investigación incluyen solo a personas que desean ser parte de ellos. Le pedimos, que por favor se tome su tiempo para decidir si participará, y discutir su decisión con su familia, amigos, con su profesional de la salud mental, o su médico si lo desea. Si tiene alguna pregunta hágasela a las investigadoras.

Se les está invitando a usted y a su hijo a ser parte del estudio porque su hijo presenta problemas de atención, de conducta, académicos y/o sociales en la escuela.

### ¿Porqué se está realizando este estudio?

El propósito de este estudio es aprender acerca de la eficacia de un programa entre escuela y hogar en línea para mejorar la atención y la conducta de estudiantes en México: CLS-FUERTE. El programa incluye un componente de habilidades parentales, un componente de orientación a los profesores de aula, y un componente de construcción de habilidades de los niños. Los resultados que surjan de este estudio promoverán más investigaciones de intervenciones efectivas y el entrenamiento de personal escolar para mejorar la atención y la conducta de los niños/as.

# ¿Quién paga el estudio?

Este estudio está financiado por una premio federal del Instituto Nacional de Salud, ganado por las Dras. Lauren Haack y Eva Araujo.

# ¿Cuántas personas formarán parte del estudio?

Un total de 88 estudiantes, sus padres/familiares, y personal clínico escolar de 11 escuelas participarán en este estudio

# ¿Qué pasará si mi hijo y yo formamos parte del estudio?

Si usted está de acuerdo en participar, y el maestro/a de su hijo también está de acuerdo en participar, el siguiente procedimiento sucederá:

- 1. Primero, realizaremos procedimientos de selección para confirmar que usted y su hijo pueden participar en el programa. Usted da el consentimiento a su escuela y a nuestro *staff* del programa para compartir información confidencial sobre su hijo, y consentimiento para que la maestra/o de su hijo responda instrumentos/cuestionarios del programa. La selección que es requerida para el estudio, consiste en lo siguiente:
  - Usted y la maestra/o de su hijo responderán los cuestionarios sobre la conducta de su hijo/a.
  - Si, basándonos en estos cuestionarios, su hijo cumple con los criterios del estudio, usted y la maestra de su hijo responderán cuestionarios acerca del funcionamiento de su hijo.

Si todos los criterios se cumplen, su hijo será elegido para continuar en el estudio; si los criterios no se cumplen se le pedirá a la escuela que le ofrezca otro tipo de opciones de ayuda. La información que hasta el momento se ha recabado por los investigadores, se quedará con ellos, para que sean reportadas las características de las familias que no participaron en este estudio.

- 2. Después, usted, su hijo y la maestra del niño participarán en un programa en línea (remoto) vía videoconferencia, que consiste en los siguientes componentes:
  - O Un componente de maestros, el cual consiste en una orientación grupal de maestros de 60 minutos y dos reuniones de seguimiento de 20-30 minutos con los maestros, el personal clínico escolar, los padres y los niños en un periodo de 6 semanas. Durante estas reuniones, diseñaremos y revisaremos adaptaciones en la clase de su niño para su mejora. Un sistema de anotaciones entre escuela-hogar llevaremos a cabo para mantener y premiar la conducta de su hijo.
  - O Un componente de padres, el cual consiste en seis sesiones grupales de 90 minutos con los padres en un periodo de 6 semanas. Estas sesiones se enfocaran en estrategias que ayudarán a su hijo a funcionar mejor en la casa, escuela, y con sus pares, así como a mejorar la calidad de la relación familiar. Los padres aplicarán estrategias dando instrucción, usando premios y consecuencias, y estableciendo rutinas y esquemas de organización para ayudar al manejo de la conducta de su hijo. En el último grupo se realizará una sesión con los niños y los padres para celebrar y alentar la participación de los niños y su éxito en el programa. Todos los cuidadores de cualquiera de los niños que participan podrán asistir a la sesión de grupo.
  - Un componente de niños que consiste en seis sesiones de 40 a 60 minutos, durante ese tiempo su hijo participará en sesiones de entrenamiento de habilidades con otros niños. Estos grupos serán durante los horarios de clase o justo después de clases..
- 3. Usted, el maestro de su hijo y el personal clínico escolar, completarán instrumentos sobre fiabilidad y aceptabilidad del programa, se responderán durante y después del programa. Además, después del programa, usted y el maestro de su hijo responderán de nuevo los cuestionarios acerca del funcionamiento del niño También invitaremos a todos los participantes a otorgar retroalimentación acerca de su experiencia con el programa en grupos focales y entrevistas.

# ¿Se realizarán video y audio grabaciones durante el estudio?

Todas las sesiones de grupo serán video-grabadas usando una plataforma de videoconferencia segura (e.g. zoom). Estas sesiones serán grabadas digitalmente y estarán resguardadas en un servidor de base de datos seguro para ser revisados después por los clínicos/investigadores, con el fin de evaluar las reuniones y

Caretaker Consent Form 

para propósitos de investigación y entrenamiento. Las grabaciones serán resguardas en nuestro sistema protegido con contraseña en la página web del entrenamiento del programa Colaborativo para Habilidades de la Vida en línea (CLS-Remote), usando una cuenta privada de video-streaming en un programa como Vimeo. Las grabaciones serán identificadas solo con números, y ninguno de sus nombres aparecerán en ellas. Las grabaciones serán guardadas indefinidamente para propósitos de investigación y entrenamiento, y desarrollo de los objetivos. La grabación es necesaria para entrenamientos, análisis y desarrollo de la investigación.

# ¿Qué sucede si su hijo está tomando medicamento para TDAH?

Si su hijo está tomando medicamento, sigue siendo elegible para el presente proyecto siempre y cuando esté tomando la misma dosis de medicamente los meses anteriores (justo antes de la selección). Su hijo puede continuar con su medicación mientras participe en el presente proyecto.

### Lugar del estudio

Todos los procedimientos del estudio se llevarán a cabo en línea o en la escuela de su hijo.

# ¿Cuánto tiempo estaremos mi hijo y yo en el estudio?

El tiempo total será obligatorio para todas las familias participantes, también el llenado de las escalas de medición durante el programa (una al inicio del estudio, y una al final del programa). Estas evaluaciones toman entre 1 y 2 horas. La participación en el programa incluye asistir durante seis semanas a reuniones grupales de padres de 90 minutos, seis semanas de grupos de niños de 40-60 minutos, y una reunión entre padres, maestros, personal clínico escolar y niños de 20-30 minutos.

# ¿Podemos mi hijo y yo dejar de participar en el estudio?

Si. Usted, o su hijo, pueden decidir no participar en cualquier momento. Solo dígaselo a algún miembro del equipo del estudio cuando lo desee.

También, los investigadores del estudio pueden detener la participación de usted o su hijo si se considera que no le interesa, o que no sigue las reglas del estudio, o si el estudio se detiene.

# ¿Qué riesgos podemos tener mi hijo o yo en el estudio?

- Potenciales riesgos al responder los cuestionarios: Los riesgos que incluyen son que algunas
  personas pueden sentirse incómodas al ser entrevistados, observador, o cuando responden
  cuestionarios sobre aspectos personales. Para prevenir estos riesgos se cuenta con un personal
  capacitado, incluyendo psicólogos infantiles. Los cuestionarios y el programa serán llevados acabo
  por profesionales de la salud mental con experiencia que han sido entrenados de forma cuidadosa
  sobre los sentimientos y el bienestar de los participantes.
- Potenciales riesgos en grupos en línea: Como parte de la participación en este programa, los participantes estarán en grupos virtuales donde se incluye la interacción con a otros padres y niños, y donde compartirán información personal con otras familias que tengan problemas similares. Esto puede ser vergonzoso o juzgado por algunas familias. Sin embargo, la experiencia y la satisfacción de los participantes de otros estudios que hemos realizado con el mismo tipo de grupos ha sido positiva. Todos los padres y niños participantes serán instruidos acerca de la confidencialidad y se les pedirá que no revelen la identidad de ningún miembro del grupo, ni repitan información personal de otros miembros del grupo. Para evitar este tipo de riesgo se cuenta con un personal altamente capacitado y

Caretaker Consent Form 

psicólogos infantiles disponibles; todo el personal estará entrenado en proteger la identidad de la información.

- Potenciales riesgos de ser grabados: Los principales riesgos incluyen que algunas personas se sienten incómodas cuando son grabadas. La pérdida de la confidencialidad es el mayor riesgo si la identidad de los niños es accidentalmente descubierta por alguien más que vea o escuche la grabación; este es menor riesgo en las audio grabaciones que en los videos. Las grabaciones en video y audio durante las sesiones de padres, maestros y niños serán usadas solo para investigación y propósitos de entrenamiento del estudio, y se mantendrán bajo llave en un gabinete en el cubículo de investigación durante el estudio y después de su término. Las grabaciones serán etiquetadas sólo con números; las etiquetas no incluyen nombres.
- Para más información sobre los riesgos, por favor pregunte a alguno de los investigadores.

# ¿Hay algún beneficio por formar parte del estudio?

Puede no haber beneficios directos para usted o su hijo al participar en el estudio. No podemos prometer que usted o su hijo recibirán algún beneficio personal de la participación de este estudio. Este estudio dará un seguimiento cuidadoso de la conducta de su hijo. Los beneficios principales que pueden derivarse pueden ser la reducción de los problemas de atención y/o conducta de su hijo, y una mejora en lo académico y sus relaciones sociales como resultado de la participación en la intervención. También tendrá el beneficio educativo de participar en un experimento científico y saber más acerca de su hijo a partir de la evaluación.

# ¿Qué otras opciones tengo si no quiero formar parte del estudio?

Las otras opciones pudieran incluir no formar parte de este estudio de investigación, tener una intervención normal y/o que los problemas de conducta no sean tomados en cuenta en un estudio, o formar parte de otro estudio. Si usted decide no participar en este estudio, no habrá ninguna amonestación. Su decisión no afecta el cuidado de su hijo o el trato que se le da en la escuela.

# ¿Qué información sobre mi persona y sobre mi hijo se mantendrá en privado?

La participación en investigaciones incluye perder privacidad. Haremos todo lo posible por asegurarnos de que la información personal adquirida en este estudio permanezca en privado. Sin embargo, no podemos garantizar total privacidad. Su información personal puede ser usada si es requerida por la ley. Algunas organizaciones revisan nuestros registros de investigación para que la calidad esté garantizada incluyendo el Instituto Nacional de Salud o el Comité de Recursos Humanos de UCSF.

La información acerca de usted y su hijo se mantendrá como confidencial lo más posible. Ni su nombre ni el de su hijo será usado en algún reporte de publicación acerca de este estudio. Todos los registros se identificarán sólo con un código numérico, y los registros permanecerán guardados en servidor de base de datos seguro. Hay algunas circunstancias especiales que pueden provocar quebrantar la confidencialidad. Esas circunstancias consisten en (a) suicidio, o intento o plan de homicidio de alguno de los miembros de la familia, o (b) abuso del niño. Todos los miembros del grupo de investigación está entrenado para registrar o notificar de manera inmediata al Investigador Principal (PI) si descubre alguna de esas circunstancias (a) o (b), estar junto a cualquiera de los participantes si este se encuentra en peligro hasta que tenga un cuidado apropiado. El PI evaluará la situación y realizará los pasos necesarios para resolver el riesgo, incluyendo dar atención de emergencia, advertir de cualquier víctima potencial, dando intervención en crisis, o haciendo un reporte de abuso a los servicios de protección infantil.

Caretaker Consent Form 

# ¿Cuál es el costo al formar parte del estudio?

No se le cobrará a usted (ni a su seguro personal en caso de tenerlo) por ninguno de los procedimientos del estudio.

# ¿Me pagarán por ser parte del estudio?

Se le pagarán \$200.00 pesos cada vez que complete los cuestionarios (antes y después del programa), siendo un total de \$400.00 pesos.

# ¿Quién puede responder mis dudas sobre el estudio?

Si usted tiene alguna pregunta, comentario o preocupación sobre su participación en el estudio, debería hablar con los investigadores. Puede contactar a la Dra. Araujo al número (667) 798-93-85. Si por alguna razón usted no desea hacer esto, o si sigue teniendo dudas o preocupaciones después de hablar con la Dra. Araujo, puede contactar al Comité de Ética de la Universidad Autónoma de Sinaloa, quienes se encargan de la protección de los voluntarios en los proyectos de investigación. También puede contactar a este comité en caso de tener dudas sobre sus derechos como participante de una investigación.

Puede encontrar en el siguiente link: <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> una descripción del programa, tal como es solicitado por las leyes de Estados Unidos. Esta página de internet no incluye información de su identificación personal. Sin embargo, dicha página si incluirá un resumen de los resultados de este estudio. Puede usted acceder a esta página cuando lo desee.

#### CONSENTIMIENTO

Usted tendrá una copia de este consentimiento para que la tenga consigo. La persona que firma a continuación es quien le ha explicado toda esta información y respondido a sus preguntas.

LA PARTICIPACIÓN EN LA INVESTIGACIÓN ES VOLUNTARIA. Usted o su hijo tienen el derecho de negar ser parte del estudio, o retirarse en cualquier momento sin alguna multa o pérdida de beneficios a los que tiene derecho.

| Si usted desea p | articipar junto con su hijo en este estudio, por favor firme debajo. |
|---|---|
| Fecha | Firma del padre para consentimiento |
| | Nombre del padre (impreso) |
| Fecha | Persona que obtiene el consentimiento |
| | o, usted da permiso para que su hijo sea incluido en este estudio. Su permiso es necesario considerando que su hijo y no puede dar consentimiento por sí mismo. |
| Fecha | Padre o Tutor Legal |

Caretaker Consent Form 

### CONSENTIMIENTO PARA PARTICIPAR EN ESTUDIO DE INVESTIGACIÓN

Programa Escuela-Hogar en línea para mejorar la atención y la conducta de estudiantes mexicanos

Para niños de 5 a 12 años de edad

### ¿Porqué nos estamos reuniendo con usted?

Queremos informarte acerca de algo que estamos realizando y que llamamos Estudio de Investigación. Un estudio de investigación es cuando diferentes doctores recolectan suficiente información para aprender más acerca de algo que ocurre. La Dra. Eva Araujo y algunos otros doctores están realizando un estudio para aprender más sobre cómo ayudar a los niños a tener más amigos y mejorar en la escuela. Después de explicarte más acerca de ello, te preguntaremos si deseas participar o no en este estudio.

### ¿Porqué estamos realizando este estudio?

Estamos realizando este estudio para buscar más formas de ayudar a los niños. Esperamos aprender más acerca de las diversas cosas que pueden ayudar a los niños a mejorar en la escuela y llevarse mejor con otros niños y con su familia. En todo el estudio, habrá 88 niños y sus familias.

### ¿Qué pasará si acepto participar en el estudio?

Si estás de acuerdo en participar en este estudio, esto es lo que pasará:

Te haremos algunas preguntas a ti y a los maestros acerca de cómo te llevas en la casa, la escuela y con tus amigos.

Después, sea durante el otoño o la primavera de este año escolar, que será decidido al azar (como una moneda al aire), estarás en un grupo con otros niños de la escuela. Aprenderá formas de llevarte mejor con otros niños, jugarás algunos juegos, y aprenderás a tener la tarea lista. El grupo será muy divertido. También te reunirás con tus papás y maestros para que les muestres todo lo que habrás aprendido en el grupo.

### ¿Alguna cosa del estudio te dañará?

Nada en el estudio daña. Te sentirás cómodo respondiendo las preguntas, pero tus respuestas podrán ayudar a saber cómo los niños se llevan con sus padres y con otros niños.

### ¿Serás mejor si participas en el estudio?

No podemos estar seguros de eso. Quizás no seas mejor. O, quizás mejores bastante en la escuela y en cómo te llevas con tu familia y amigos.

# ¿Tienes alguna pregunta?

Puedes preguntar lo que quieras en cualquier momento. Puedes preguntar ahora mismo. O puedes preguntar después. Puedes hablarme a mí o a alguien más.

# ¿Tienes que estar en el estudio?

No. Nadie se molestará si tu no quieres estar en el estudio. Si no quieres estar en el estudio solo dínoslo. O si quieres estar en el estudio, dilo. Y, recuerda, puedes decir si ahora, y después cambiar de opinión. Es tu decisión.

Si no quieres participar en este estudio, solo dilo. Si quieres participar en este estudio, por favor di "Si, si quiero participar en el estudio".

Tu familia tendrá una copia de este documento para que tú lo tengas.

# FIRMA DE LA PERSONA QUE DISCUTIÓ EL CONSENTIMIENTO

| He explicado el estudio a | (nombre del niño/a) en un lenguaje |
|---|---|
| que él/ella puede entender, y el/la niño/a acordó de form | |
| Firma de la persona que discutió el consentimiento | Fecha |
| Nombre de la persona que discutió el consentimiento (im | ppresa) |